CLINICAL TRIAL: NCT04770922
Title: Pharmacogenomic Analysis of 6-mercaptopurine in Pediatric Acute Lymphoblastic Leukemia
Brief Title: Pharmacogenomic Analysis in Pediatric Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Cipherome, Inc. (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: C04-001
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric; Adverse Drug Event
Keywords: adverse drug event; acute lymphoblastic leukemia; mercaptopurine; pharmacogenomics
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Observational study of previously collected biobank specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric ALL patients on 6-mercaptopurine: Pediatric ALL patients treated with 6-mercaptopurine who did not experience neutropenia.
- Pediatric ALL patients on 6-mercaptopurine with neutropenia: Pediatric ALL patients treated with 6-mercaptopurine who experienced neutropenia.

SUMMARY:
This is a retrospective biobank study evaluating the impact of novel genetic variants in a population of 6-mercaptopurine treated pediatric acute lymphoblastic leukemia patients.

DETAILED DESCRIPTION:
The study objective is to clinically validate that the presence of recently discovered novel genetic variation adversely affects a population of 6-mercaptopurine treated pediatric acute lymphoblastic leukemia patients using biobank samples.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric acute lymphoblastic leukemia (ALL) subjects
* Received 6-mercaptopurine
* Available biobank (bone marrow or blood) sample(s) from which deoxyribonucleic acid (DNA) can be extracted
* White blood cell (WBC) levels

Exclusion Criteria:

* Pediatric ALL subjects who did NOT receive 6-mercaptopurine
* No biobank sample
* No WBC level

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population are pediatric patients, under 21 years of age, diagnosed with acute lymphoblastic leukemia patients between April 20, 2012 to August 6, 2020, and received 6-mercaptopurine for therapeutic purposes. All patients were recruited by the investigators at Stanford University Lucile Packard Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Novel genetic variants impact on 6-mercaptopurine adverse drug reactions | 1 year
  Objective is to clinically validate the presence of novel genetic variants and its impact on adverse drug reactions in a population of pediatric ALL patients treated with 6-MP

SECONDARY OUTCOMES:
Evaluating relationship of genetic variants to ancestry | 1 year
  A secondary objective of this study is to compare the impact of the novel genetic variants with other known genetic variants contributing to ADR risk.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Sakamoto, MD, PhD, Principal Investigator — Stanford University; Stephanie M Smith, MD, Study Director — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bhatia S, Landier W, Hageman L, Chen Y, Kim H, Sun CL, Kornegay N, Evans WE, Angiolillo AL, Bostrom B, Casillas J, Lew G, Maloney KW, Mascarenhas L, Ritchey AK, Termuhlen AM, Carroll WL, Wong FL, Relling MV. Systemic Exposure to Thiopurines and Risk of Relapse in Children With Acute Lymphoblastic Leukemia: A Children's Oncology Group Study. JAMA Oncol. 2015 Jun;1(3):287-95. doi: 10.1001/jamaoncol.2015.0245. PMID 26181173
- [Background] Park Y, Kim H, Choi JY, Yun S, Min BJ, Seo ME, Im HJ, Kang HJ, Kim JH. Star Allele-Based Haplotyping versus Gene-Wise Variant Burden Scoring for Predicting 6-Mercaptopurine Intolerance in Pediatric Acute Lymphoblastic Leukemia Patients. Front Pharmacol. 2019 Jun 11;10:654. doi: 10.3389/fphar.2019.00654. eCollection 2019. PMID 31244663
- [Result] Relling MV, Gardner EE, Sandborn WJ, Schmiegelow K, Pui CH, Yee SW, Stein CM, Carrillo M, Evans WE, Klein TE; Clinical Pharmacogenetics Implementation Consortium. Clinical Pharmacogenetics Implementation Consortium guidelines for thiopurine methyltransferase genotype and thiopurine dosing. Clin Pharmacol Ther. 2011 Mar;89(3):387-91. doi: 10.1038/clpt.2010.320. Epub 2011 Jan 26. PMID 21270794
- [Result] Yang JJ, Landier W, Yang W, Liu C, Hageman L, Cheng C, Pei D, Chen Y, Crews KR, Kornegay N, Wong FL, Evans WE, Pui CH, Bhatia S, Relling MV. Inherited NUDT15 variant is a genetic determinant of mercaptopurine intolerance in children with acute lymphoblastic leukemia. J Clin Oncol. 2015 Apr 10;33(11):1235-42. doi: 10.1200/JCO.2014.59.4671. Epub 2015 Jan 26. PMID 25624441
- [Result] Lennard L. Implementation of TPMT testing. Br J Clin Pharmacol. 2014 Apr;77(4):704-14. doi: 10.1111/bcp.12226. PMID 23962279